CLINICAL TRIAL: NCT06291220
Title: A Phase 1 Study Evaluating Safety, Pharmacokinetics, and Efficacy of ABBV-453 in Adult Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Brief Title: A Study Assessing Adverse Event and How Oral ABBV-453 Moves Through the Body in Adult Participants With Relapsed or Refractory (R/R) Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Acronym: 453 Ph1 CLL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-291; 2023-507637-19 (Other: EU CT)
Record Dates: First submitted 2024-02-27; First posted 2024-03-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Chronic Lymphocytic Leukemia: Small Lymphocytic Lymphoma; SLL; CLL; ABBV-453
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Part A: Cohort 1.1 ABBV-453 Dose A (Experimental): Participants will receive obinutuzumab during the debulking period followed escalating doses of ABBV-453, until the dose A is achieved, during the 5 year study duration.
  Interventions: Drug: Obinutuzumab; Drug: ABBV-453

INTERVENTIONS:
Drug: Obinutuzumab — Intravenous Infusion
Drug: ABBV-453 — Oral; Tablet

SUMMARY:
Chronic lymphocytic leukemia (CLL) is the most common leukemia in Western countries. The purpose of this study is to assess how well ABBV-453 works adult participants with relapsed/refractory (R/R) untreated CLL/small lymphocytic lymphoma (SLL). Adverse events, pharmacokinetics, and change in disease activity will be assessed.

ABBV-453 is an investigational drug for the treatment of CLL and SLL. Participants will be enrolled with a specific target dose and receive obinutuzumab during the debulking period followed escalating doses of ABBV-453, until the appropriate target dose is achieved. Approximately 60 adult participants with previously R/R CLL/SLL will be enrolled in the study in approximately 40 sites across the world.

Participants will receive intravenous (IV) obinutuzumab as part of the debulking period, followed by escalating doses of oral ABBV-453 until the appropriate target dose is achieved. The estimated study duration is 3 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory (R/R) chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL) that has received at least 2 prior systemic therapies and have no available (or established) therapies known to provide clinical benefit and to which the participant would consent to receiving.
* Laboratory values meeting those listed in the protocol.

Exclusion Criteria:

* QT interval corrected for heart rate (QTc) using Fridericia's correction of > 470 msec (females) or > 450 msec (males), Grade 3 arrythmia, and/or other clinically significant cardiac abnormalities.
* Known to be B-cell leukemia/lymphoma 2 inhibitor (BCL-2i) refractory or has received a BCL-2i-containing regimen within (6 months) of starting study drug (e.g., venetoclax, lisaftoclax, BGV-11417).
* Has active human immunodeficiency virus (HIV) infection. HIV testing is not required unless required locally.
* Recent history (within 6 months) of:

  * Congestive heart failure (defined as New York Heart Association, Class 2 or higher).
  * Ischemic cardiovascular event.
  * Cardiac arrhythmia requiring pharmacological or surgical intervention.
  * Pericardial effusion.
  * Pericarditis.
* Consumes known moderate or strong inhibitors of cytochrome P450 3A isoform subfamily (CYP3A) within 14 day or 5 half-lives of the drug (whichever is shorter) before the first dose of ABBV-453.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to 3 Years
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Maximum Administered Dose (MAD) of ABBV-453 | Up to 18 Months
  MAD is defined as the highest administered dose if no maximum tolerated dose (MTD) is determined.
Maximum Tolerated Dose (MTD) of ABBV-453 | Up to 18 Months
  MTD is defined as the highest dose administered that does not result in a final determination of de-escalate at that dose level.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ABBV-453 | Up to 30 Months
  Cmax is defined as the maximum observed plasma/serum concentration of ABBV-453.
Time to Maximum Observed Concentration (Tmax) of ABBV-453 | Up to 30 Months
  Tmax is defined as the time to maximum observed concentration of ABBV-453.
Area Under the Plasma/Serum Concentration Versus Time Curve (AUC) of ABBV-453 | Up to 30 Months
  Area under the plasma/serum concentration versus time curve (AUC) of ABBV-453.
Overall Response Rate (ORR) | Up to 3 Years
  Percentage of participants achieving a complete response (CR), complete response with incomplete count recovery (CRi), partial response (PR), or nodular partial response (nPR) using disease-specific criteria per the International Workshop on Chronic Lymphocytic Leukemia (iwCLL, 2018).
Duration of Response (DOR) for Participants with PR/nPR or Better | Up to 3 Years
  DOR is defined as the time between the initial PR or better response assessment per Investigator according to iwCLL criteria to the time of progressive disease (PD) or death of any cause, whichever occurs earlier.
Complete response rate (CRR) | Up to 3 Years
  CRR is defined as the percentage of participants with a best overall response (BOR) of CR or CRi per Investigator review according to iwCLL for participants with relapsed or refractory CLL/SLL, regardless of reasons for study drug discontinuation, and prior to start of subsequent anti-cancer therapies in the participants receiving at least one dose of ABBV-453 monotherapy.
Duration of Complete Response (DOCR) | Up to 3 Years
  DOCR is defined as the time between the initial CR/CRi response assessment per Investigator according to iwCLL criteria to the time of PD or death of any cause, whichever occurs earlier.
Percentage of Participants Achieving an Minimal Residual Disease (MRD) Negativity Among Participants Achieving a PR, nPR, CR, or CRi | Up to 3 Years
  MRD response is defined as < 1 cell in 10,000 leukocytes (< 10^-4).
Progression-free survival (PFS) | Up to 3 Years
  PFS is defined as time from first study treatment to a documented PD (based on iwCLL criteria) as determined by the Investigator, or death due to any cause, whichever occurs earlier.
Overall survival (OS) | Up to 3 Years
  OS is defined as the time from the first date of study treatment until date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (21):
- United States (6):
  - City of Hope /ID# 253904, Duarte, California
  - City of Hope - Orange County Lennar Foundation Cancer Center /ID# 267158, Irvine, California
  - Intermountain Health St. Vincent Regional Hospital - Cancer Centers of Montana /ID# 264622, Billings, Montana
  - Atrium Health /ID# 265136, Charlotte, North Carolina
  - Duplicate_Duke Cancer Center /ID# 258707, Durham, North Carolina
  - MD Anderson Cancer Center /ID# 253713, Houston, Texas
- Australia (4):
  - Royal Prince Alfred Hospital /ID# 263129, Sydney, New South Wales
  - Gold coast University Hospital /ID# 255785, Southport, Queensland
  - Austin Health /ID# 256776, Heidelberg, Victoria
  - Royal Perth Hospital /ID# 256464, Perth, Western Australia
- Germany (5):
  - Universitaetsklinikum Ulm /ID# 263148, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Halle (Saale) /ID# 263299, Halle, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel /ID# 263150, Kiel, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin /ID# 263433, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 263730, Hamburg
- Israel (3):
  - Yitzhak Shamir Medical Center /ID# 257626, Ẕerifin, Central District
  - Hadassah Medical Center-Hebrew University /ID# 254721, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 254383, Ramat Gan, Tel Aviv
- Italy (3):
  - IRCCS Ospedale San Raffaele /ID# 263064, Milan, Milano
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 263065, Bologna
  - Azienda Ospedaliera di Perugia - Ospedale S. Maria della Misericordia /ID# 263062, Perugia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-291